CLINICAL TRIAL: NCT03998930
Title: Brain-computer Interface in the Diagnosis of Disorders of Consciousness
Brief Title: Evaluation of Consciousness by Brain-computer Interface in Severely Brain Damaged Patients
Acronym: AWAKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: M2H laboratory, Montpellier University (Other); IMT Mines Alès, Alès, France (Unknown); University Hospital, Montpellier (Other); Hôpital d'Uzès, Uzès, France (Unknown); Clinique Fontfroide, Montpellier, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Local/2017/FF-02; 2017-A02539-44 (Other: ANSM)
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Traumatic Brain Injury With Prolonged Loss of Consciousness; Stroke; Brain Hypoxia
Keywords: Disorders of consciousness,; Brain Computer Interface; P300; Motor imagery
MeSH Terms: conditions — Stroke; Hypoxia, Brain; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- brain injuried patients (Experimental): * Clinical evaluation of consciousness by the Coma Recovery Scale Revised (CRS-R),
  * 15-minute break between the two evaluations.
  * Paraclinical evaluation of consciousness by the brain-machine interface by measuring evoked potentials P300 auditory and vibrotactile and recording the EEG signal during a motor imaging task (imagine moving the right or left wrist).
  Interventions: Other: Clinical evaluation of consciousness by the Coma Recovery Scale Revised (CRS-R)

INTERVENTIONS:
Other: Clinical evaluation of consciousness by the Coma Recovery Scale Revised (CRS-R) — Paraclinical evaluation of consciousness by the brain-machine interface by measuring evoked potentials P300 auditory and vibrotactile and recording the EEG signal during a motor imaging task
  Other Names: other

SUMMARY:
The objective of this study is to show that the measurement of auditory and vibro-tactile evoked potentials, or the recording of the EEG signal during a motor imaging task, can be used in routine clinical situations to explore the state of consciousness of subjects in Non-responsive Awakening (or Chronic Vegetative State) or in Minimal Consciousness (or relational state) after a severe brain injury.

Assumptions :

* Correlation between patient response rates obtained with the brain-machine interface and their clinical consciousness score (Coma Recovery Scale Revised score)
* Differentiation of the parameters of the evoked potentials P300 between patients in a vegetative state and those in a state of minimal consciousness

DETAILED DESCRIPTION:
this is a pilot study on information obtained using a medical device marketed in accordance with CE standards, multicentric and prospective.

The study participation consists of five assessments of the subjects' level of awareness. Each evaluation lasts a total of two hours.

Patients will be assessed in their rooms as follows:

* Clinical evaluation of consciousness by the Coma Recovery Scale Revised (CRS-R), a clinical scale considered as the "gold-standard". Duration 45 minutes (standard care in routine care)
* 15-minute break between the two evaluations.
* Paraclinical evaluation of consciousness by the brain-machine interface by measuring evoked potentials P300 auditory and vibrotactile and recording the EEG signal during a motor imaging task (imagine moving the right or left wrist). Duration 60 minutes.

Instructions are given to the subject via headphones, in French. For the analysis of the evoked potentials, vibrotactile stimuli are delivered to the wrists and ankle of the subject. For auditory evoked potentials, auditory stimuli are delivered by headphones. The volume can be changed.

These assessments that we will perform with the brain-machine interface are similar to the assessments and stimulation of awakening and awareness sessions performed by speech-language pathologists in the departments concerned (presentation of visual and auditory stimuli). CRS-R is used in routine care to assess patients' level of consciousness. There is no recommendation on the type of additional examination to be performed (neuroimaging, EEG, evoked potentials) or on their frequency for the evaluation of patients' consciousness at a distance from their initial brain injury.

Evaluation by the brain-machine interface in the room makes it possible to avoid transport to the complementary examination services (Medical Imaging Services, Neurological Functional Explorations) which cause fatigue (patient whose vigilance is fluctuating) which can make the complementary examination non-contributory. Patients are also not assessed at a date and time set by a complementary examination service and room assessment allows the patient to be assessed in the best conditions for him/her when he/she appears to be at his/her highest level of consciousness and rested (after consultation with the family and/or healthcare team).

Total duration of each session of a maximum of 2 hours, including the installation and uninstallation of the brain-machine interface.

Patients receive their usual treatment and continue to participate in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* The patient and/or his/her trusted person, relative or legal representative must have given free and informed consent and signed the consent
* The patient must be a member or beneficiary of a health insurance plan
* The patient is available for a 10-day follow-up
* Women and men are included
* The patient is at least 18 years old
* Subjects with conscious disorder, non-respondents after traumatic brain injury (head injury) or non-traumatic brain injury (hemorrhagic and/or ischemic stroke, cerebral anoxia, encephalitis).

Exclusion Criteria:

* Subject is participating in another intervention study
* The subject is in an exclusion period determined by a previous study
* The subject or his or her trusted person, relative or legal representative refuses to sign the consent
* The patient is pregnant or breastfeeding
* The subject has hemodynamic, respiratory and/or neurological instability
* The subject has an ENT infection in the ears (wearing headphones)
* History of auditory and/or sensory sensory impairment
* Psychiatric history (other than anxiety-depressive syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
correlation between the response of patients obtained with the brain-machine interface (detection of auditory and vibrotactile P300 and modifications of EEG signal during a motor imagery task) and their clinical consciousness score | Inclusion
  correlation coefficient (units: -1; 1)
correlation between the response of patients obtained with the brain-machine interface (detection of auditory and vibrotactile P300 and modifications of EEG signal during a motor imagery task) and their clinical consciousness score | Day 2
  correlation coefficient (units: -1; 1)
correlation between the response of patients obtained with the brain-machine interface (detection of auditory and vibrotactile P300 and modifications of EEG signal during a motor imagery task) and their clinical consciousness score | Day 4
  correlation coefficient (units: -1; 1)
correlation between the response of patients obtained with the brain-machine interface (detection of auditory and vibrotactile P300 and modifications of EEG signal during a motor imagery task) and their clinical consciousness score | Day 6
  correlation coefficient (units: -1; 1)
correlation between the response of patients obtained with the brain-machine interface (detection of auditory and vibrotactile P300 and modifications of EEG signal during a motor imagery task) and their clinical consciousness score | Day 10
  correlation coefficient (units: -1; 1)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Montpellier, Montpellier
  - Clinique Fontfroide, Montpellier
  - CHU de Nîmes, Nîmes
  - Hôpital d'Uzès, Uzès

IPD SHARING:
Plan to Share IPD: No